CLINICAL TRIAL: NCT03776331
Title: Characterization of Vascular Functions in Myeloma Patients Before and During Anti-tumor Therapy
Brief Title: Vascular Functions in Myeloma Patients During Anti-tumor Therapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Fadi Al-Rashid, Principal Investigator, University Hospital, Essen
Other Study IDs: Vascular-Myelom
Record Dates: First submitted 2018-11-10; First posted 2018-12-14 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Cardiooncology; Myeloma; Endothelial Dysfunction
Keywords: Myeloma; Flow mediated dilation; Endothelial Dysfunction; Proteasome inhibitors
MeSH Terms: conditions — Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Myeloma Patients
  Interventions: Diagnostic Test: Flow mediated dilation
- Controll group
  Interventions: Diagnostic Test: Flow mediated dilation

INTERVENTIONS:
Diagnostic Test: Flow mediated dilation — Measurement of the change in the vasodilatative reserve of the brachial artery

SUMMARY:
Treatment options for multiple myeloma have increased significantly over the last years with the approval of immunomodulatory drugs (IMiDs) and proteasome inhibitors (PIs). These therapies have markedly improved overall survival for these patients to a median of 5-7 years. Due to the advanced age, the myeloma patient collective has a high prevalence of pre-existing cardiovascular comorbidities. In addition, the primary disease process contributes to cardiovascular complications. With the beginning of anti-tumor therapy, an increased incidence of cardiovascular complications in myeloma patients can be determined. This includes hypertension, left ventricular dysfunction, heart failure and both arterial and venous thromboembolic events. The detailed mechanism by which proteasome inhibitors and immunomodulatory agents lead to increased cardiovascular events is not established at this time. Endothelial dysfunction, as a possible mechanism of cardiovascular toxicity, is difficult to assess. Flow-mediated dilation (FMD) is an noninvasive method to measure endothelial function by assessing the change in the vasodilatative reserve of the brachial artery. Several independent recent investigations implicate that vascular (endothelial) dysfunction precedes hypertension and heart failure. This has been related to a reduced level of metabolites of the l-arginine-nitric oxide (NO) signaling pathway.

Hypothesis:

1. Anti-myeloma therapy exert vascular toxicity by limiting endothelial function. Endothelial function, assessed by the change in the vasodilatative reserve of the brachial artery (flow-mediated dilation = FMD) decreases after myeloma therapy.
2. Patients with multiple myeloma have a limited endothelial function compared to a healthy control group.

A total of 40 myeloma patients will be examined. Measurements will be taken at baseline, 1 month and 6 month after myeloma therapy. Patients should not have received chemotherapy for at least 3 months. Furthermore a healthy sex- and age-matched control group will be examined.

DETAILED DESCRIPTION:
Treatment options for multiple myeloma have increased significantly over the last years with the approval of immunomodulatory drugs (IMiDs) and proteasome inhibitors (PIs). These therapies have markedly improved overall survival for these patients to a median of 5-7 years, many continue to live for more than 10 years. Due to the advanced age, the myeloma patient collective has a high prevalence of pre-existing cardiovascular comorbidities. In addition, the primary disease process contributes to cardiovascular complications. With the beginning of anti-tumor therapy, an increased incidence of cardiovascular complications in myeloma patients can be determined. This includes hypertension, left ventricular dysfunction, heart failure and both arterial and venous thromboembolic events.

Proteasome inhibitors including bortezomib and carfilzomib, and immunomodulatory agents, e.g. lenalidomide, represent cornerstone therapies for multiple myeloma. The most common therapy choices are Bortezomib-based therapy (VCD, VC) and Carfilzomib-based therapy (KRD, KD). Induction therapy is given 4-6 cycles followed by autologous hematopoietic cell transplantation. Thereafter, many patients receive consolidation therapy. In patients not eligible for autologous hematopoietic cell transplantation, a prolonged course of initial chemotherapy is typically administered. The proteasome inhibitor Bortezomib is used predominately in the front line setting, while second-generation carfilzomib is used in relapsed/refractory disease.

Despite their efficacy, increased rates of cardiovascular complications occur in patients exposed to these particular therapies. Higher incidences of cardiac adverse events including hypertension, arrhythmia, heart failure, ischemic heart disease and cardiomyopathy has been reported in patients receiving carfilzomib and bortezomib. Immunomodulatory agents are known to increase the risk of venous thromboembolic disease particularly when combined with dexamethasone or other chemotherapy. Furthermore, increased incidence of myocardial infarction (MI) and cerebrovascular events has been demonstrated in patients treated with lenalidomide. The mechanism of PI- and IMiD-associated cardiotoxicity is not fully elucidated. PIs inhibit proteasome activity, leading to the accumulation of abnormal proteins which in turn activates apoptotic pathways in myeloma cells. IMiDs bind cereblon, a component of the E3 ubiquitin ligase which promotes proteasome-mediated degradation of the transcription factors, IKZF1 and IKZF. It is unclear if the protein degradation properties of these drugs contribute to cardiotoxicity, although clinical features of the toxicity suggest endothelial cell injury and dysfunction. It is possible that CV events may be augmented when these two classes of medications are co-administered and further enhanced by the additional endothelial stress conferred by steroids. The detailed mechanism by which proteasome inhibitors and immunomodulatory agents lead to increased cardiovascular events is not established at this time.

Endothelial dysfunction, as a possible mechanism of cardiovascular toxicity, is difficult to assess. Flow-mediated dilation (FMD) is an noninvasive method to measure endothelial function by assessing the change in the vasodilatative reserve of the brachial artery. Several independent recent investigations implicate that vascular (endothelial) dysfunction precedes hypertension and heart failure. This has been related to a reduced level of metabolites of the l-arginine-nitric oxide (NO) signaling pathway.

Hypothesis:

1. Anti-myeloma therapy exert vascular toxicity by limiting endothelial function. Endothelial function, assessed by the change in the vasodilatative reserve of the brachial artery (flow-mediated dilation = FMD) decreases after myeloma therapy.
2. Patients with multiple myeloma have a limited endothelial function compared to a healthy control group.

Study design:

A total of 40 myeloma patients will be examined. Measurements will be taken at baseline, 1 month 6 month after myeloma therapy. Patients should not have received chemotherapy for at least 3 months. Furthermore a healthy sex- and age-matched control group will be examined.

Primary endpoint:

• Endothelial function, assessed by the change in the vasodilatative reserve of the brachial artery (flow-mediated dilation = FMD), between baseline and 1 month data

Secondary endpoints:

* Endothelial function, assessed by the vasodilatative reserve of the brachial artery (flow-mediated dilation = FMD) between baseline data in myeloma patients and control group
* Change of left ventricular pump function (3D-EF, global longitudinal strain)
* Alteration of echocardiographic parameters of diastolic dysfunction
* Change in dyspnea symptoms (NYHA Classification)
* Modification of cardiac biomarkers (NT-pro BNP, Troponin)
* Change of circulating NO-Pool
* Change in metabolomics (Biobank)
* Change in arterial stiffness and augmentation index
* Change of quality of life rated according to Medical Outcomes Short-Form Survey, SF-36, Minnesota Living With Heart Failure Questionnaire
* Change in blood pressure

ELIGIBILITY:
Included in the study are myeloma patients with planned bortezomib, carfilzomib and lenalidomide-based chemotherapy and 20 subjects from a healthy normal population.

Inclusion Criteria:

* Age ≥ 18 years
* written consent

Exclusion Criteria:

* Severe pulmonary, valvular, or congenital heart disease with clinical dyspnoea symptoms
* Life expectancy less than 6 months
* Unstable angina pectoris or indication for coronary revascularization
* Valvular disease (aortic valve and mitral regurgitation greater than moderate, and aortic valve or mitral valve stenosis greater than moderate)
* Atrial fibrillation or flutter
* Chronic renal insufficiency (Cockcroft-Gault GFR <30 mL / min)
* Severe cirrhosis (Child-Pugh B and C)
* Current or future indication for therapy with organic nitrates
* Leading non-cardiac cause of clinical dyspnea symptoms, such as high-grade obesity or lung disease in need of glucocorticoid therapy or oxygen therapy
* Other cause of clinical dyspnea symptoms, such as high-grade obesity or lung disease with need for glucocorticoid therapy or oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cohorts will be selected of the population of patients of the university clinic of Essen
Sampling Method: Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2018-12-28 (Estimated); Primary Completion 2019-12-28 (Estimated); Study Completion 2020-03-28 (Estimated)

PRIMARY OUTCOMES:
Change of endothelial function, assessed by the change in the vasodilatative reserve of the brachial artery (flow-mediated dilation = FMD) | between baseline and 1 month data

SECONDARY OUTCOMES:
Change of endothelial function, assessed by the change in the vasodilatative reserve of the brachial artery (flow-mediated dilation = FMD) | between baseline and 6 month data
Change of endothelial function, assessed by the change in the vasodilatative reserve of the brachial artery (flow-mediated dilation = FMD) | between 1 and 6 month data
Change of endothelial function, assessed by the vasodilatative reserve of the brachial artery (flow-mediated dilation = FMD) between baseline data in myeloma patients and control group | baseline data
Change of left ventricular pump function (3D-EF) | between baseline and 1 month data/baseline and 6 month data/1 and 6 month data
Change of left ventricular pump function (global longitudinal strain) | between baseline and 1 month data/baseline and 6 month data/1 and 6 month data
Alteration of grade of diastolic dysfunction | between baseline and 1 month data/baseline and 6 month data/1 and 6 month data
  Assesed by E, E/A, E/e', IVRT, DT, e', e'/a', TEI index, sPAP, according to ASE/EACVI GUIDELINES AND STANDARDS, Recommendations for the Evaluation of Left Ventricular Diastolic Function by Echocardiography: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging, Sherif et al, 2016, J Am Soc Echocardiogr, 2016
Change in dyspnea symptoms (NYHA Classification) | between baseline and 1 month data/baseline and 6 month data/1 and 6 month data
Change in concentration of Troponin | between baseline and 1 month data/baseline and 6 month data/1 and 6 month data
Change in concentration of NT-pro BNP | between baseline and 1 month data/baseline and 6 month data/1 and 6 month data
Change in circulating arginine-nitric oxide (NO) metabolites | between baseline and 1 month data/baseline and 6 month data/1 and 6 month data
  Levels of arginine, citrulline, ornithine, asymmetric dimethylarginine (ADMA), symmetric dimethylarginine (SDMA), and N-monomethylarginine (MMA)
Change in levels of circulating arginine | between baseline and 1 month data/baseline and 6 month data/1 and 6 month data
Change in leves of circulating citrulline | between baseline and 1 month data/baseline and 6 month data/1 and 6 month data
Change in levels of circulating ornithine | between baseline and 1 month data/baseline and 6 month data/1 and 6 month data
Change in levels of circulating asymmetric dimethylarginine (ADMA) | between baseline and 1 month data/baseline and 6 month data/1 and 6 month data
Change in levels of circulating symmetric dimethylarginine (SDMA) | between baseline and 1 month data/baseline and 6 month data/1 and 6 month data
Change in levels of circulating N-monomethylarginine (MMA) | between baseline and 1 month data/baseline and 6 month data/1 and 6 month data
Change in pulse wave velocity as a parameter of arterial stiffness | between baseline and 1 month data/baseline and 6 month data/1 and 6 month data
Change in augmentation index | between baseline and 1 month data/baseline and 6 month data/1 and 6 month data
  Augmentation index (AIx), the pressure difference between the shoulder on the pressure wave and systolic pressure expressed as a ratio of pulse pressure is widely used as a proxy of wave reflection
Change of quality of life rated according to Minnesota Living With Heart Failure Questionnaire | between baseline and 1 month data/baseline and 6 month data/1 and 6 month data
  The questionnaire is comprised of 21 important physical, emotional and socioeconomic ways heart failure can adversely affect a patient's life. After receiving brief standardized instructions, the patient marks a 0 (zero) to 5 scale to indicate how much each itemized adverse of heart failure has prevented the patient from living as he or she wanted to live during the past 4 weeks. The questionnaire is simply scored by summation of all 21 responses.
Change of quality of life rated according to Medical Outcomes Short-Form Survey | between baseline and 1 month data/baseline and 6 month data/1 and 6 month data
  The SF-36 consists of 36 questions and is a general health questionnaire that provides information about the health status of the patient through 8 different dimensions. He makes statements about:
  General Health Perception, Physical Health, Restricted physical role function, Physical pain, Vitality, Mental Healt, Restricted emotional role function, Social functioning. For the evaluation of the SF-36 questionnaire v1.0 you first recode all answers in predefined points using a recoding table. Then you calculate the average score of all questions of the respective health dimension, e.g. physical health, so you have 8 average points for the 8 dimensions. These 8 scores now describe the health status of the patient in their respective dimensions, which can then be assessed using comparison charts.
  The possible score ranges from 0 to 100 points. 0 points represent the greatest possible restriction of health, while 100 points represent the absence of health restrictions.
Change in blood pressure (systolic, diastolic and MAD) | between baseline and 1 month data/baseline and 6 month data/1 and 6 month data

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Totzeck, Principal Investigator — Universitätsklinikum Essen AOeR

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR